CLINICAL TRIAL: NCT03902132
Title: Effects of Core Stability Exercises on Lower Back Pain and Quality of Life in Post-menopausal Women.
Brief Title: Core Muscle Stability on Low Back Pain and Quality of Life in Post- Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Sumaira Kanwal
Record Dates: First submitted 2019-03-20; First posted 2019-04-03 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Backache, Low
Keywords: Backache; Core Stability exercises; Post menopausal
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: Single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Stability exercises group (Experimental): Core Stability exercises
  Interventions: Other: Core Stability exercises group
- Traditional low back physical therapy group (Active Comparator): Traditional low back physical therapy management
  Interventions: Other: Traditional low back physical therapy group

INTERVENTIONS:
Other: Core Stability exercises group — Core Stability Exercises were given in addition to the traditional physical therapy treatment as given to the control group. It included moist heat pack (10mins), Transcutaneous Electrical Nerve Stimulation (10 min), and strengthening regimen (2 sets with 15 isometric repetitions each).
  Arms: Core Stability exercises group
Other: Traditional low back physical therapy group — The control group was given traditional low backache physical therapy management such as moist heat pack, TENS, and strengthening regimen (2 sets with 15 isometric repetitions each)
  Arms: Traditional low back physical therapy group

SUMMARY:
Low back pain, postural dysfunction, loss of balance control and stability are musculoskeletal changes that occur over life span due to aging process and are inevitable. Core stability exercises are an effective means to counteract these changes.The study was executed with initially n=35 subjects selected as per proposal, but only n=24 subjects completed the study with n=14 in experimental group and n=10 in control group. Experimental group received core stability exercises and control group received conventional physical therapy treatment for 12 weeks. Baseline assessment was done, then at 6 week and again at end of intervention.Following outcome measures were used in study Numeric pain rating scale (NPRS), Utain quality of life (UQOL), Oswestry disability index (ODI), manual muscle testing (MMT) flexion and extension. Data was analysed using Statistical package for social sciences SPSS- 21.

DETAILED DESCRIPTION:
About total of 80% of population once in their life have gone through Low back pain that cause significant loss of productive working hours along with disability. People suffering from chronic low back pain and impaired function, often experience anxiety, depression, as well as effects on work and social life. Low back pain largely effects the women population, aged 45-60 years, accounting for distress on a social as well as economic level.

Age predicted incidence of low back pain (LBP) was also found to be higher in post-menopausal women. (90% between 40 and 60, mean age 50.1 years). Decline in psychological and cognitive function along with other health related conditions like heart disease, mood swings, risk of cancer are of particular importance in post-menopausal women affecting their quality of life.

The hormonal changes occurring in women during and after menopause, may also have an impact on health-related quality of life (HRQoL) particularly at the physical, psychological, and sexual spheres. Physical therapy remains the most advanced conservative option for the treatment of LBP Core stability or core strengthening exercises are increasingly becoming an important element of the sports world of therapeutics as it provides distal mobility with proximal stability(9). Core stability and strengthening exercises are supported strongly by theoretical principles for the treatment of spinal disorders that helps in decreasing pain and improving function in people suffering from LBP.

Core strengthening has attracted limited research attention so far yet it has been promoted as a mode of rehabilitation, for performance enhancement and as preventive measure of injuries related to the musculoskeletal and lumbar spine. The significance of core stability exercises in postmenopausal women with backache has been overlooked so far. The proposed study focused on Core stability exercises in Postmenopausal woman with Lower back pain to investigate the effects of core strength training on lower back pain, disability, strength and the quality of life in postmenopausal woman.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-60 years
* Post menopausal women
* Having low back pain (NPRS >2)

Exclusion Criteria:

* Participants with physical or mental illness making them unable to participate in the study

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Post menopausal women
Enrollment: 24 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | The score were recorded at baseline, at the (6th week) and at 12th visit (12th week) to determine the reduction or aggravation of pain followed by treatment in both control and experimental groups.
  Changes from the Baseline, NPRS was used to measure the patient's pain intensity and divided from 0-11 into 11 divisions. 0 means absence of pain. 1 to 3 demonstrates mild degree of pain. 4 to 6 moderate level of pain and 7 to 10 means severe degree of pain. Patients were directed to select a number that best described the pain at the moment.
Utian Quality of Life (UQOL): | The score were recorded at baseline, at the 6th visit (6th week) and at 12th visit (12th week) followed by treatment in both control and experimental groups.
  Changes from the Baseline, Quality of life (QOL), a statistical outcome variable must be measured in a regulatory trial research in a clinical care settings. Utian QOL scale (UQOL) is dynamically based on sensitivity of well-being as distinct from menopausal symptoms.

SECONDARY OUTCOMES:
Oswestry disability Index (ODI): | The score were recorded at baseline, at 6th session the (6th week) and at 12th visit (12th week) followed by treatment in both control and experimental groups.
  Changes from the Baseline, ODI is an effective tool to provide information on the extent of backache affecting the patient ability to cope with tasks of everyday life. Ten sections are included in the ODI tool with a total possible score of 5 for each section. The first statement carries a score of 0, and the last has a score of 5.
Manual Muscle Testing (MMT) | The score were recorded at baseline, at the (6th week) and at 12th visit (12th week) followed by treatment in both control and experimental groups.
  Changes from the Baseline, MMT of flexors and extensors. It consists of 0- 5 grades. 0 indicates no visible or palpable contraction, 1 indicates Visible or palpable contraction with no motion, 2 indicates full range of motion (ROM) with gravity eliminated, 3 full range of motion anti gravity, 4 shows Full ROM against gravity, moderate resistance, 5 indicates Full ROM against gravity, maximal resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Irum Yaqoob, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Imran Amjad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmed R, Shakil-Ur-Rehman S, Sibtain F. Comparison between Specific Lumber Mobilization and Core-Stability Exercises with Core-Stability Exercises Alone in Mechanical low back pain. Pak J Med Sci. 2014 Jan;30(1):157-60. doi: 10.12669/pjms.301.4424. PMID 24639852
- [Background] Kamper SJ, Apeldoorn AT, Chiarotto A, Smeets RJ, Ostelo RW, Guzman J, van Tulder MW. Multidisciplinary biopsychosocial rehabilitation for chronic low back pain: Cochrane systematic review and meta-analysis. BMJ. 2015 Feb 18;350:h444. doi: 10.1136/bmj.h444. PMID 25694111
- [Background] Kozinoga M, Majchrzycki M, Piotrowska S. Low back pain in women before and after menopause. Prz Menopauzalny. 2015 Sep;14(3):203-7. doi: 10.5114/pm.2015.54347. Epub 2015 Sep 30. PMID 26528111
- [Background] Park JJ, Shin J, Youn Y, Champagne C, Jin E, Hong S, Jung K, Lee S, Yeom S. Bone mineral density, body mass index, postmenopausal period and outcomes of low back pain treatment in Korean postmenopausal women. Eur Spine J. 2010 Nov;19(11):1942-7. doi: 10.1007/s00586-010-1559-7. Epub 2010 Sep 1. PMID 20811756
- [Background] Dalal PK, Agarwal M. Postmenopausal syndrome. Indian J Psychiatry. 2015 Jul;57(Suppl 2):S222-32. doi: 10.4103/0019-5545.161483. PMID 26330639
- [Background] Moratalla-Cecilia N, Soriano-Maldonado A, Ruiz-Cabello P, Fernandez MM, Gregorio-Arenas E, Aranda P, Aparicio VA. Association of physical fitness with health-related quality of life in early postmenopause. Qual Life Res. 2016 Oct;25(10):2675-2681. doi: 10.1007/s11136-016-1294-6. Epub 2016 Apr 16. PMID 27085340
- [Background] Akuthota V, Ferreiro A, Moore T, Fredericson M. Core stability exercise principles. Curr Sports Med Rep. 2008 Feb;7(1):39-44. doi: 10.1097/01.CSMR.0000308663.13278.69. PMID 18296944
- [Background] Thompson PD, Buchner D, Pina IL, Balady GJ, Williams MA, Marcus BH, Berra K, Blair SN, Costa F, Franklin B, Fletcher GF, Gordon NF, Pate RR, Rodriguez BL, Yancey AK, Wenger NK; American Heart Association Council on Clinical Cardiology Subcommittee on Exercise, Rehabilitation, and Prevention; American Heart Association Council on Nutrition, Physical Activity, and Metabolism Subcommittee on Physical Activity. Exercise and physical activity in the prevention and treatment of atherosclerotic cardiovascular disease: a statement from the Council on Clinical Cardiology (Subcommittee on Exercise, Rehabilitation, and Prevention) and the Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity). Circulation. 2003 Jun 24;107(24):3109-16. doi: 10.1161/01.CIR.0000075572.40158.77. No abstract available. PMID 12821592
- [Background] Akuthota V, Nadler SF. Core strengthening. Arch Phys Med Rehabil. 2004 Mar;85(3 Suppl 1):S86-92. doi: 10.1053/j.apmr.2003.12.005. PMID 15034861